CLINICAL TRIAL: NCT02552251
Title: Comparative Study of the Use of Glucocorticoids in the Treatment of Congenital Adrenal Hyperplasia in Its Classical Form
Brief Title: COrticosteroid in Congenital Adrenal Hyperplasia
Acronym: COCA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11-059
Record Dates: First submitted 2015-07-27; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: hydrocortisone (Experimental): hydrocortisone equivalent to physiological doses for each patient Strategy: administration of glucocorticoids during sequences of eight weeks
  Interventions: Biological: Hormonal balance measurements; Biological: metabolic balance measurements; Biological: bone balance measurements; Behavioral: quality of life assessment
- B :dexamethasone (DECTANCYL) (Experimental): dexamethasone equivalent to physiological doses for each patient Strategy: administration of glucocorticoids during sequences of eight weeks
  Interventions: Biological: Hormonal balance measurements; Biological: metabolic balance measurements; Biological: bone balance measurements; Behavioral: quality of life assessment
- C : prednisone (CORTANCYL) (Experimental): prednisone equivalent to physiological doses for each patient Strategy: administration of glucocorticoids during sequences of eight weeks
  Interventions: Biological: Hormonal balance measurements; Biological: metabolic balance measurements; Biological: bone balance measurements; Behavioral: quality of life assessment

INTERVENTIONS:
Biological: Hormonal balance measurements
Biological: metabolic balance measurements
Biological: bone balance measurements
Behavioral: quality of life assessment

SUMMARY:
Congenital adrenal hyperplasia (CAH) results from a deficiency of a key enzyme in the biosynthesis of cortisol, mainly 21-hydroxylase, resulting in its classic form a neonatal salt loss syndrome and / or a virilization syndrome in girls. The treatment of the disorder in adulthood involves administering steroidal compounds with the aim to substitute the gluco- and mineralocorticoid deficit on the one hand, and effectively curb the adrenal hyperplasia and adrenal androgen pathway in girls . The terms of glucocorticoid treatment are not clearly codified and are based on several steroidal compounds and various protocols. The advantages in terms of adrenal suppression and disadvantages - including bone and metabolic - different treatments have not been clearly established in the literature. The main objective of this study is to compare among adults with HCS in its classical form the impact on hormonal parameters adrenal suppression glucocorticoid of 3 types of treatment administered to equivalent dose and according to the usual procedures. The secondary objective is to compare in the same patients the impact of different drugs and treatments on several metabolic bone parameters. The study will include 40 adult patients bearing a HCS in its classical form and will include 3 treatment sequences of eight weeks each, during which they will be administered sequentially in random order at random and according to the known equivalences hydrocortisone, prednisone (CORTANCYL) and dexamethasone (DECTANCYL).

Randomization will be stratified based on previous DMARDs in the investigation that may be different for different patients, knowing that France hydrocortisone and dexamethasone are used mainly for the treatment of congenital adrenal hyperplasia. The judging criteria will be: i) the criteria of adrenal hormone suppression: plasma levels of testosterone, androstenedione, 17 OHP, ACTH and diurnal variations of the 17 OH progesterone salivary ii) the criteria of the metabolic impact of glucocorticoids: plasma glucose levels , blood lipids, and insulin sensitivity index HOMA-R calculated from glucose and insulin, iii) the criteria of bone impact of glucocorticoids: plasma for CTX bone resorption and bone alkaline phosphatase P1NP for bone formation iv) the living quality criteria evaluated by the PGWB Questionnaire (Psychological General Well-Being). The duration of the study period will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Pubescent women over 18 in genital activity (premenopausal)
* Suffering from congenital adrenal hyperplasia in its classical form with salt loss or pure virilizing
* Patients who have presented signs of congenital adrenal hyperplasia in its classical form (salt wasting syndrome and / or neonatal masculinization) with elevation of 17 OH progesterone with diagnosis of enzyme block 21 hydroxylase.
* Patients currently treated by: 1 or 2 Oral compound glucocorticoid as replacement and suppressive therapy + 1 mineralocorticoid if necessary with effective control of substitution + possibly by estrogen-progestin pill.

Exclusion Criteria:

* Liver disease, kidney, bone, diabetes, severe dyslipidemia, pregnancy
* Postmenopausal women, age over 55 years
* Concomitant therapy: glucocorticoids supra-physiological doses for other indications, bisphosphonates, vitamin D, oral antidiabetic agents or insulin, lipid lowering agents (eg inflammatory disease, asthma, systemic disease ... ..).
* participation of the subject to another biomedical research protocol for this study
* Inability to submit to medical monitoring study for geographical, social or psychological.
* Severe calorie diet planned or carried out during the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
hormonal parameters | change over baseline, week 8, week 16, week 24
  6 points salivary 17 OHP cycle, and 8 am plasma ACTH,testosterone and androstenedione

SECONDARY OUTCOMES:
parameters of bone turnover: | change over baseline, week 8, week 16, week 24
  CTX and bone alkaline phosphatase P1NP
metabolic parameters: | change over baseline, week 8, week 16, week 24
  blood glucose and insulin, cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol
Quality of Life | change over baseline, week 8, week 16, week 24
  Psychological General Well-Being questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Service Endocrinologie et Maladies Métaboliques, Caen, France